CLINICAL TRIAL: NCT02114788
Title: INTERACTIVE SECTIONS OF AN INTERNET-BASED INTERVENTION INCREASE PATIENT EMPOWERMENT: A RANDOMIZED CONTROLLED STUDY WITH CHRONIC BACK PAIN PATIENTS
Brief Title: Interactive Sections Of An Internet-Based Intervention Increase Patient Empowerment: A Study With Chronic Back Pain Patients
Status: Completed | Type: Observational
Sponsor: University of Lugano (Other)
Responsible Party: Principal Investigator, Silvia Riva, Dr, University of Lugano
Other Study IDs: FNS100013_130030/1
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Group 1 (Control): Access to a Static Version of the Website Containing Only Static Features (i.e. Library, First Aid, and FAQ); Group2 (Intervention) Access to an Interactive Version of the Website Containing Both Static and Interactive Features

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- group 1: No intervention
- Group 2: Intervention with interactive website
  Interventions: Other: Internet-based

INTERVENTIONS:
Other: Internet-based
  Groups: Group 2

SUMMARY:
The aim of the study is to study how to improve patients' management of chronic back pain, particularly their management of prescription medication, through increasing health literacy and patient empowerment through an internet based intervention. We do this by designing both patient education materials and physician communication strategies to increase literacy and volitional components of patients. We will test two conditions using a website called Oneself: one providing only information (literacy-only control) and a second providing relational communications designed to increase both literacy and volitional empowerment. To test the self-management enhancing effects of empowerment and health literacy, we will conduct a longitudinal experiment with 51 chronich back pain patients over two months. This span of time is the minimum necessary to achieve a systematic change in self-management and literacy skills, increasing also the range of possible decisions to be made and actions to be real-ized by the patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged > 18 years,
2. having suffered from back pain for at least 3 months,
3. no concurrent involvement in other studies.

Exclusion Criteria:

1. No access/limited access to computer and internet
2. concurrent diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are screened through their healthcare provider at selected clinics and rehabilitation centers in the Canton Ticino (Switzerland).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Empowerment level (psychological measure) | 8 weeks
  Empowerment is a pychological outcome measure. Patient empowerment is defined as a complex construct that includes different individual competencies and skills. Empowerment can be considered a multilevel and multidimensional construct closely linked to self-determination and self-efficacy.
  Empowerment is measured the with the Psychological Empowerment Scale According to the scale, empowerment is a multidimensional concept composed of four cognitive dimensions (or task assessments): impact (or the degree to which behavior is seen as "making a difference"), competence (or the degree to which a person can perform task activities skillfully), meaningfulness (or the individual's intrinsic caring about a given task), and choice (or whether a person's behavior is perceived as self-determined).

SECONDARY OUTCOMES:
Medication misuse Physical exercise Pain burden | 8 weeks
  Medication misuse is measured with the Prescription Medication Use and Perception of Risk Instrument. The scale is scored as a continuous measure to provide greater sensitivity ranging from 0 (strongly disagree) to 6 (strongly agree) with higher scores indicating greater level of medication misuse.
  Physical exercise in leisure time is measured with the respective sub-dimensions from the Short Questionnaire to Assess Health-Enhancing Physical Activity and it gives the amount of time spent in physical exercise in hours/week
  Pain burden is measured with six items from the Chronic Pain Grading Scale that gives two measures related with pain: pain disability perception and pain intensity perception

CONTACTS AND LOCATIONS:
Locations (1):
- Insitute of Communication nad Health, University of Lugano, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Riva S, Camerini AL, Allam A, Schulz PJ. Interactive sections of an Internet-based intervention increase empowerment of chronic back pain patients: randomized controlled trial. J Med Internet Res. 2014 Aug 13;16(8):e180. doi: 10.2196/jmir.3474. PMID 25119374
- See also: website used for the study — http://www.oneself.ch